CLINICAL TRIAL: NCT01757678
Title: HeartFlowNXT - HeartFlow Analysis of Coronary Blood Flow Using Coronary CT Angiography: NeXt sTeps
Brief Title: HeartFlowNXT - HeartFlow Analysis of Coronary Blood Flow Using Coronary CT Angiography
Acronym: HFNXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HeartFlow, Inc. (Industry)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: CP-902-001
Record Dates: First submitted 2012-12-18; First posted 2012-12-31 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease Computed Fractional Flow Reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: prospective, multicenter study to evaluate the diagnostic performance of cCTA plus FFRCT employing ≥64-detector row CT scanners for the detection and exclusion of significant obstructive CAD, as defined by invasively-measured FFR, the reference standard
Masking Description: No Masking
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard of care: FFR, ICA, cCTA, FFRct (Other): (ICA) Invasive coronary angiography with (FFR) fractional flow reserve measurement in standard of care environment, and cCTA (computed coronary tomography angiography) and FFRct Analysis (fractional flow reserve computed tomography)
  Interventions: Procedure: ICA (Invasive Coronary Angiography); Procedure: FFR (Fractional Flow Reserve); Procedure: cCTA (coronary computed tomography angiography); Other: FFRct Analysis (Fractional Flow Reserve Computed Tomography)

INTERVENTIONS:
Procedure: ICA (Invasive Coronary Angiography) — Per the protocol, patients will have an Invasive Coronary Angiography.
Procedure: FFR (Fractional Flow Reserve) — Per the protocol, patients will have a Fractional Flow Reserve procedure.
Procedure: cCTA (coronary computed tomography angiography) — Per the protocol, patients will have a coronary computed tomography angiography.
Other: FFRct Analysis (Fractional Flow Reserve Computed Tomography) — Per the protocol, patients will have a fractional flow reserve computed tomography.

SUMMARY:
To determine the diagnostic performance of FFRCT by coronary computed tomographic angiography (cCTA), as compared to cCTA alone, for non-invasive determination of the presence of a hemodynamically significant coronary lesion, using direct measurement of fractional flow reserve (FFR) during cardiac catheterization as a reference standard.

DETAILED DESCRIPTION:
Recently, coronary Computed Tomography Angiography (cCTA) of 64-detector rows or greater has emerged as a novel non-invasive imaging modality that is capable of providing high-resolution images of coronary artery lesions (Budoff 2008; Miller 2008; Meijboom 2008). While cCTA demonstrates good diagnostic performance for detection and exclusion of anatomic coronary artery stenoses, numerous prior studies have revealed an unreliable relationship between detection of obstructive anatomic coronary artery stenoses by cCTA and hemodynamically (HD)-significant coronary artery disease (CAD), identified by myocardial perfusion SPECT or fractional flow reserve (FFR) (Di Carli 2007; Klauss 2007; Rispler 2007; van Werkhoven 2009). Individual subjects may have HD-significant CAD despite cCTA assessment demonstrating angiographically mild (<50%) maximal stenosis (Schuijf 2006). These findings emphasize the need for additional measures beyond anatomic stenosis severity for the detection and exclusion of HD-significant CAD.

Measurement of FFR during invasive cardiac catheterization represents the "gold standard" for assessment of the hemodynamic significance of coronary artery lesions (Kern 2010). Anatomic coronary artery stenosis assessment by quantitative coronary angiography (QCA) also correlates very poorly with FFR Melikian 2010). This was highlighted by the results of the FAME study in which FFR-guided coronary revascularization improved healthcare and economic outcomes compared to the conventional angiographically guided strategy (Pijls 2010; Tonino 2009; Tonino 2010).

The major disadvantage of FFR is that it has to be measured invasively. HeartFlow, Inc. ('HeartFlow') has recently developed a non-invasive method to determine FFR which computes the hemodynamic significance of CAD (FFRCT) from subject-specific cCTA data using computational fluid dynamics under rest and simulated maximal coronary hyperemic conditions. Preliminary results in subjects suggest that FFRCT accurately predicts the hemodynamic significance of coronary lesions when compared to directly-measured FFR during invasive cardiac catheterization (Koo 2011).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Subject providing written informed consent
* Scheduled to undergo a clinically indicated Invasive Coronary Angiogram (ICA)
* Has had ≥64 multidetector row cCTA within 60 days prior to ICA or agrees to undergo cCTA with ≥64 multidetector row cCTA within 60 days prior to ICA

Exclusion Criteria:

* Percutaneous coronary intervention (PCI) has been performed any time prior to ICA.
* Prior coronary artery bypass graft (CABG) surgery
* Contraindication to beta blocker agents, nitrates, or adenosine, including 2nd or 3rd degree heart block; sick sinus syndrome; long QT syndrome; severe hypotension; severe asthma, severe COPD or bronchodilator-dependent COPD
* Suspicion of acute coronary syndrome (acute myocardial infarction and unstable angina)
* Recent prior myocardial infarction within 30 days prior to cCTA or between cCTA and ICA
* Known complex congenital heart disease
* Prior pacemaker or internal defibrillator lead implantation
* Prosthetic heart valve
* Tachycardia or significant arrhythmia
* Impaired chronic renal function (serum creatinine >1.5 mg/dl)
* Subjects with known anaphylactic allergy to iodinated contrast
* Pregnancy or unknown pregnancy status in subject of childbearing potential
* Body mass index >35 at time of cCTA
* Subject requires an emergent procedure
* Evidence of ongoing or active clinical instability, including acute chest pain (sudden onset), cardiogenic shock, unstable blood pressure with systolic blood pressure <90 mmHg, and severe congestive heart failure (NYHA III or IV) or acute pulmonary edema
* Any active, serious, life-threatening disease with a life expectancy of less than 2 months
* Inability to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bjarne Norgaard, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Ihdayhid AR, Norgaard BL, Gaur S, Leipsic J, Nerlekar N, Osawa K, Miyoshi T, Jensen JM, Kimura T, Shiomi H, Erglis A, Jegere S, Oldroyd KG, Botker HE, Seneviratne SK, Achenbach S, Ko BS. Prognostic Value and Risk Continuum of Noninvasive Fractional Flow Reserve Derived from Coronary CT Angiography. Radiology. 2019 Aug;292(2):343-351. doi: 10.1148/radiol.2019182264. Epub 2019 Jun 11. PMID 31184558
- [Derived] Ovrehus KA, Gaur S, Leipsic J, Jensen JM, Dey D, Botker HE, Ahmadi A, Achenbach S, Ko B, Norgaard BL. CT-based total vessel plaque analyses improves prediction of hemodynamic significance lesions as assessed by fractional flow reserve in patients with stable angina pectoris. J Cardiovasc Comput Tomogr. 2018 Jul-Aug;12(4):344-349. doi: 10.1016/j.jcct.2018.04.008. Epub 2018 May 8. PMID 29866619
- [Derived] Ko BS, Wong DT, Norgaard BL, Leong DP, Cameron JD, Gaur S, Marwan M, Achenbach S, Kuribayashi S, Kimura T, Meredith IT, Seneviratne SK. Diagnostic Performance of Transluminal Attenuation Gradient and Noninvasive Fractional Flow Reserve Derived from 320-Detector Row CT Angiography to Diagnose Hemodynamically Significant Coronary Stenosis: An NXT Substudy. Radiology. 2016 Apr;279(1):75-83. doi: 10.1148/radiol.2015150383. Epub 2015 Oct 6. PMID 26444662
- [Derived] Norgaard BL, Leipsic J, Gaur S, Seneviratne S, Ko BS, Ito H, Jensen JM, Mauri L, De Bruyne B, Bezerra H, Osawa K, Marwan M, Naber C, Erglis A, Park SJ, Christiansen EH, Kaltoft A, Lassen JF, Botker HE, Achenbach S; NXT Trial Study Group. Diagnostic performance of noninvasive fractional flow reserve derived from coronary computed tomography angiography in suspected coronary artery disease: the NXT trial (Analysis of Coronary Blood Flow Using CT Angiography: Next Steps). J Am Coll Cardiol. 2014 Apr 1;63(12):1145-1155. doi: 10.1016/j.jacc.2013.11.043. Epub 2014 Jan 30. PMID 24486266
- [Derived] Gaur S, Achenbach S, Leipsic J, Mauri L, Bezerra HG, Jensen JM, Botker HE, Lassen JF, Norgaard BL. Rationale and design of the HeartFlowNXT (HeartFlow analysis of coronary blood flow using CT angiography: NeXt sTeps) study. J Cardiovasc Comput Tomogr. 2013 Sep-Oct;7(5):279-88. doi: 10.1016/j.jcct.2013.09.003. Epub 2013 Oct 1. PMID 24268114

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: FFR and ICA: Single arm
  Measured FFR: Fractional Flow Reserve
Period: Overall Study
Arm/Group | Standard of Care: FFR and ICA
Started | 276
Completed | 276
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: FFR and ICA: Single arm
  Measured FFR (Fractional Flow Reserve) and ICA (Invasive Coronary Angiography)
Arm/Group | Standard of Care: FFR and ICA
Number analyzed (Participants) | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 175
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 91
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 179
  More than one race | 0
  Unknown or Not Reported | 6
Diabetes [Number; unit: participants]
  With Diabetes | 62
  Without Diabetes | 214
Hypertension [Number; unit: participants]
  With Hypertension | 188
  Without Hypertension | 88
Hyperlipidemia [Number; unit: participants]
  With Hyperlipidemia | 214
  Without Hyperlipidemia | 60
  Unknown Hiperlipidemia Status | 2
Current smoker [Number; unit: participants]
  Current Smoker | 50
  Former Smoker | 106
  Never Smoked | 118
  Unknown | 2
Previous myocardial infarction [Number; unit: participants]
  Previous Myocardial Infarction | 5
  No Previous Myocardial Infarction | 271
Body Mass Index, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 26 (4)
Creatinine, mg/dl [Mean (Standard Deviation); unit: mg/dl] | 0.9 (.2)
Left ventricular ejection fraction, % [Mean (Standard Deviation); unit: percent] | 62 (7)

OUTCOME MEASURES:

1. Secondary Outcome: AUC of FFRct Versus Coronary CTA for Demonstration of Ischemia (≤0.80) on a Per-vessel Basis
Time Frame: 1 day
Population: 22 of the 276 enrolled subjects were excluded by the FFR/QCA Core Lab, leaving an ITD population of 254 subjects. 3 additional subjects were excluded from the ITD analysis due to missing cCTA 30%-90% stenosis by coronary CTA.
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: Vessels
Arm/Group | FFRct vs. FFR | cCTA vs. FFR
Number analyzed (Participants) | 251 | 251
Number analyzed (Vessels) | 484 | 484
probability | .93 [0.91 to 0.95] | .79 [.74 to .84]
Statistical Analysis 1: Comparison: FFRct vs. FFR vs cCTA vs. FFR; Test type: Other; Difference in Probability = .14, 95% CI 2-sided [.09 to .19]

2. Primary Outcome: AUC of FFRct Versus Coronary CTA for Demonstration of Ischemia (≤0.80) on a Per-patient Basis
Description: The primary statistical measure will be the area under the receiver operating characteristic curve (AUC of ROC) of a patient-based model to detect hemodynamically significant obstruction. ROC graphs the change in sensitivity as the cut-point for positive/negative diagnosis moves from its lower to upper limit. FFR is used as the reference standard to determine the presence or absence of hemodynamic obstruction. For FFR, hemodynamically-significant obstruction of a coronary artery is defined as an FFR≤0.80 in any major epicardial coronary artery segment with diameter ≥2.0 mm during adenosine-mediated hyperemia. For cCTA, hemodynamically-significant obstruction of a coronary artery is defined as a stenosis >50% . FFRCT will be calculated for each patient as the minimum FFRCT in any coronary artery segment . cCTA stenosis will be calculated for each patient as the highest cCTA stenosis category for any vessel all measurements will take place only in segments with diameter ≥2.0 mm.
Time Frame: 1 day; Outcome measures were comparing FFRct to FFR. Incident time for FFR was dependent on the length of time on the cath procedure. FFRct was done remotely at HeartFlow's processing center in Redwood City with a turnaround time of 24 hours from CT scan.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: probablility
Arm/Group | FFRct vs. FFR | cCTA vs. FFR
Number analyzed (Participants) | 251 | 251
probablility | .90 [.87 to .94] | .81 [.76 to .87]
Statistical Analysis 1: Comparison: FFRct vs. FFR vs cCTA vs. FFR; Test type: Other; Difference in Probability = .09, 95% CI 2-sided [.04 to .14]

3. Secondary Outcome: Per-Patient Analysis: Diagnostic Performance of FFRct, Coronary CTA, and ICA
Time Frame: as for outcome 2
Population: 22 of the 276 enrolled subjects were excluded from the analysis by the FFR/QCA Core Lab.
Measure: Number (95% Confidence Interval); unit: percentage of tests
Groups:
- Standard of Care: FFR and ICA: (ICA) Invasive coronary angiography with (FFR) fractional flow reserve measurement in standard of care environment.
Arm/Group | Standard of Care: FFR and ICA
Number analyzed (Participants) | 254
percentage of tests
  Accuracy: ICA Stenosis >50% | 77 [71 to 82]
  Accuracy: FFRct ≤ 0.80 | 81 [76 to 85]
  Accuracy: Coronary CTA Stenosis >50% | 53 [47 to 57]
  Sensitivity: ICA Stenosis >50% | 64 [53 to 74]
  Sensitivity: FFRct ≤ 0.80 | 86 [77 to 92]
  Sensitivity: Coronary CTA Stenosis >50% | 94 [86 to 97]
  Specificity: ICA Stenosis >50% | 83 [77 to 88]
  Specificity: FFRct ≤ 0.80 | 79 [72 to 84]
  Specificity: Coronary CTA Stenosis >50% | 34 [27 to 41]
  Positive Predictive Value: ICA Stenosis >50% | 63 [52 to 73]
  Positive Predictive Value: FFRct ≤ 0.80 | 65 [56 to 74]
  Positive Predictive Value: cCTA Stenosis >50% | 40 [33 to 47]
  Negative Predictive Value: ICA Stenosis >50% | 83 [77 to 89]
  Negative Predictive Value: FFRct ≤ 0.80 | 93 [87 to 96]
  Negative Predictive Value: cCTA Stenosis >50% | 92 [83 to 97]

4. Secondary Outcome: Per Vessel Diagnostic Performance of FFRct, Coronary CTA, and ICA
Time Frame: as for outcome 2
Population: 22 of the 276 enrolled subjects were excluded from the analysis by the FFR/QCA Core Lab.
Measure: Number (95% Confidence Interval); unit: percentage of tests
Units Other Than Participants: Vessels
Arm/Group | Standard of Care: FFR and ICA
Number analyzed (Participants) | 254
Number analyzed (Vessels) | 484
percentage of tests
  Accuracy: ICA Stenosis >50% | 82 [79 to 86]
  Accuracy: FFRct ≤ 0.80 | 86 [83 to 89]
  Accuracy: Coronary CTA Stenosis >50% | 65 [61 to 69]
  Sensitivity: ICA Stenosis >50% | 55 [45 to 65]
  Sensitivity: FFRct ≤ 0.80 | 84 [75 to 89]
  Sensitivity: Coronary CTA Stenosis >50% | 83 [74 to 89]
  Specificity: ICA Stenosis >50% | 90 [86 to 93]
  Specificity: FFRct ≤ 0.80 | 86 [82 to 89]
  Specificity: Coronary CTA Stenosis >50% | 60 [56 to 65]
  Positive Predictive Value: ICA Stenosis >50% | 58 [48 to 68]
  Positive Predictive Value: FFRct ≤ 0.80 | 61 [53 to 69]
  Positive Predictive Value: cCTA Stenosis >50% | 33 [27 to 39]
  Negative Predictive Value: ICA Stenosis >50% | 88 [85 to 92]
  Negative Predictive Value: FFRct ≤ 0.80 | 95 [93 to 97]
  Negative Predictive Value: cCTA Stenosis >50% | 92 [88 to 95]

5. Post Hoc Outcome: Per-Patient Diagnostic Performance of FFRct in Patients With Intermediate Stenosis Severity (30%-70%) According to Coronary CTA
Time Frame: as for outcome 2
Population: Patients with intermediate stenosis severity (30%-70%) according to coronary CTA.
Measure: Number (95% Confidence Interval); unit: percentage of tests
Arm/Group | Standard of Care: FFR and ICA
Number analyzed (Participants) | 235
percentage of tests
  Accuracy: FFRct ≤ 0.80 | 80 [75 to 85]
  Accuracy: Coronary CTA Stenosis > 50% | 51 [44 to 57]
  Sensitivity: FFRct ≤ 0.80 | 85 [74 to 91]
  Sensitivity: Coronary CTA Stenosis >50% | 93 [85 to 97]
  Specificity: FFRct ≤ 0.80 | 79 [72 to 84]
  Specificity: Coronary CTA Stenosis > 50% | 32 [26 to 40]
  Positive Predictive Value: FFRct ≤ 0.80 | 63 [53 to 72]
  Positive Predictive Value: cCTA Stenosis > 50% | 37 [31 to 44]
  Negative Predictive Value: FFRct ≤ 0.80 | 92 [87 to 96]
  Negative Predictive Value: cCTA Stenosis > 50% | 91 [81 to 96]

ADVERSE EVENTS:
Time Frame: Index Procedure through hospital discharge
Description: Note: this study involved prospective data collection to validate in a blinded manner a non-invasive test therefore adverse event information is reported based only on the standard of care index procedure.
Groups:
- Standard of Care: ICA (Invasive Coronary Angiography): (ICA) Invasive coronary angiography in standard of care environment.
- Standard of Care: cCTA (Coronary Computed Tomography Angio): (cCTA) Coronary computed tomography angiography in standard of care environment.
- Standard of Care: FFR (Fractional Flow Reserve): (FFR) Fractional flow reserve in standard of care environment.
Arm/Group | Standard of Care: ICA (Invasive Coronary Angiography) | Standard of Care: cCTA (Coronary Computed Tomography Angio) | Standard of Care: FFR (Fractional Flow Reserve)
Serious Adverse Events (participants affected / at risk) | 5/276 | 5/276 | 5/276
Other Adverse Events (participants affected / at risk) | 53/276 | 53/276 | 53/276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care: ICA (Invasive Coronary Angiography) (N=276) | Standard of Care: cCTA (Coronary Computed Tomography Angio) (N=276) | Standard of Care: FFR (Fractional Flow Reserve) (N=276)
Coronary Dissection during invasive FFR measurement requiring percutaneous coronary intervention (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Transient cerebral ischemic attacks after ICA and invasive FFR measurement (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
Fever (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) — Fever with prolonged hospitalization
Angina Pectoris (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) — Angina pectoris following catheterization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care: ICA (Invasive Coronary Angiography) (N=276) | Standard of Care: cCTA (Coronary Computed Tomography Angio) (N=276) | Standard of Care: FFR (Fractional Flow Reserve) (N=276)
Procedural Hypotension (Injury, poisoning and procedural complications) | 9 (9) | 9 (9) | 9 (9)
Procedural Arrhythmia (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 4 (4)
Procedural Allergic Reaction (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
Procedural Angina/Chest Pain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
Procedural TIA (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
Procedural Vasovagal Response (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
Procedural Blurred Vision (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural Complete Heart Block (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural Coughing (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural Dissection (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural Distal Embolism (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural Dyspnea (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural Headache (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural Numbness (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural Perforation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural Rash/Urticaria (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural sickness during and after Adenosine (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural Vomiting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Discharge Hematoma (Injury, poisoning and procedural complications) | 9 (9) | 9 (9) | 9 (9)
Discharge Angina/Chest Pain (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 4 (4)
Discharge Headache (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 3 (3)
Discharge Arrhythmia (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
Discharge Absence Seizure (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Discharge Blurred Vision (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Discharge Chest Tightness (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Discharge Facial and Chest Rash (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Discharge Fever (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Discharge Nosebleed (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Discharge Wind Pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
13% of patients were judged to have nonevaluable cCTA images on the basis of a pre-defined image quality score. This number may be reduced with improvement of CT acquisition techniques as well a refinement of the FFRct technology.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less